CLINICAL TRIAL: NCT01859169
Title: Longterm Outcome of Photodynamic Therapy Compared With Biliary Drainage Alone in Patients With Unresectable Cholangiocarcinoma
Brief Title: Safety and Efficiency of Photodynamic Therapy for Blie Duct Carcinoma
Status: Suspended | Type: Observational
Why Stopped: Modifying the clinnicaltrials
Sponsor: li xiong (Other)
Responsible Party: Sponsor-Investigator, li xiong, Doctor（visiting staff）, Central South University
Organization: Central South University (Other)
Other Study IDs: PDT-B-01; PDT-B-01 (Other: Central South University)
Record Dates: First submitted 2013-05-10; First posted 2013-05-21 (Estimated); Last update posted 2013-05-21 (Estimated); Status verified 2013-05

CONDITIONS: Cholangiocarcinoma
Keywords: bili duct neoplasms; bile duct cancer; photodynamic therapy; biliary drainage
MeSH Terms: conditions — Cholangiocarcinoma; Bile Duct Neoplasms | interventions — Photochemotherapy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Control Group: Group that be administrated biliary drainage only
- PDT Group: Group that be administrated photodynamic therapy and biliary drainage
  Interventions: Procedure: Photodynamic therapy

INTERVENTIONS:
Procedure: Photodynamic therapy — Each patient to whom PDT was offered underwent a specific, detailed educational process by a dedicated team member(P.B., P.J., or K.E.), after which informed consent was obtained.Porfimer sodium (Photofrin; Axcan Pharma Inc, Quebec, Canada)was used as a photo sensitizing agent, administered intravenously at a dose of 2 mg/kg body weight 48 hours before illumination.A diode laser system (InGaAIP Laser Diode; Diomed Inc, An-dover, MA) with a maximum power output of 2000 mW and a wavelength of 633+-3 nm was used as a light source, delivered through a 3.0-m length fiber having a 2.5-cm-long cylindrical diffuser at its distal end (Pioneer Optics, Windsor Locks, CT).
  Groups: PDT Group

SUMMARY:
This research is a prospective randomized controlled trial.It aimed to determine longterm outcomes and factors associated with increased survival after photodynamic therapy (PDT) through T-tube compared with biliary drainage alone in patients presenting with unresectable bile duct cancer.

ELIGIBILITY:
Inclusion Criteria:

* 1.Patients with bile duct cancer 2.Patients are willing to join in this clinical trial.

Exclusion Criteria:

* 1.Patients with bile duct carcinoma can not suffer PDT procedure. 2.Allergy to photosensitizer

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with bile duct cancer
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2013-06; Primary Completion 2015-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Survival rate | one month

SECONDARY OUTCOMES:
Quality of life | one month

OTHER OUTCOMES:
Complication of therapy | one month

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Xiangya Hospital of Central South University, Changsha, Hunan, China

REFERENCES:
- [Background] Kahaleh M, Mishra R, Shami VM, Northup PG, Berg CL, Bashlor P, Jones P, Ellen K, Weiss GR, Brenin CM, Kurth BE, Rich TA, Adams RB, Yeaton P. Unresectable cholangiocarcinoma: comparison of survival in biliary stenting alone versus stenting with photodynamic therapy. Clin Gastroenterol Hepatol. 2008 Mar;6(3):290-7. doi: 10.1016/j.cgh.2007.12.004. Epub 2008 Feb 6. PMID 18255347